CLINICAL TRIAL: NCT02717585
Title: Effect of Continuous Positive Airway Pressure (CPAP) on Symptoms of Patients With Fibromyalgia Syndrome and Obstructive Sleep Apnea (OSA): A Prospective Randomized Controlled Clinical Trial
Brief Title: Effect of CPAP on Symptoms of Patients With Fibromyalgia and Obstructive Sleep Apnea
Acronym: FM-OSA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding available
Sponsor: Women's College Hospital (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-0112-B
Record Dates: First submitted 2016-03-17; First posted 2016-03-23 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Fibromyalgia; Obstructive Sleep Apnea
Keywords: Continuous Positive Airway Pressure therapy; Chronic Pain; Sleep Disturbance
MeSH Terms: conditions — Fibromyalgia; Sleep Apnea, Obstructive; Chronic Pain; Parasomnias

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): For the no intervention group (Control), patients will only receive standardized treatment for FM at the Pain Clinic. All patients will receive a multifaceted tailored regimen that incorporates one or more lines of pharmacological and/or non-pharmacological therapy. All assessment and management will be performed according to evidence-based therapeutic recommendations put forward by the Canadian Rheumatology Association and Canadian Pain Society.
- Treatment Group (CPAP) (Active Comparator): In addition to standard FM treatment at the Pain Clinic, patients who are randomized to the treatment will meet with a sleep physician for possible therapy with a Continuous Positive Airway Pressure (CPAP) machine. A CPAP titration study will be arranged for in a laboratory setting, where in addition to the regular parameters of a diagnostic sleep study, CPAP will be titrated upwards starting from 5cm H2O to an optimal setting where the obstructive respiratory events are abolished. Patients will undergo regular follow-up as determined by their sleep physician. Adherence to CPAP treatment will be recorded at follow-up visits.
  Interventions: Device: Continuous Positive Airway Pressure Therapy (CPAP)

INTERVENTIONS:
Device: Continuous Positive Airway Pressure Therapy (CPAP) — Continuous Positive Airway Pressure Therapy (CPAP) consists of a mask, fitted to the patient's face and hooked to a machine that generates positive pressure at the end of expiration to abolish obstructive apneic episodes during sleep.
  Arms: Treatment Group (CPAP)

SUMMARY:
Fibromyalgia (FM) is a chronic pain disorder associated with a wide spectrum of sleep disorders. In fact, insomnia and waking unrefreshed are currently considered part of the criteria for diagnosis. Recent studies show that sleep quality and symptoms of FM are inversely correlated. Obstructive sleep apnea (OSA) is a sleep disorder characterized by repeated episodes of complete or partial blockage of the upper airway. Nonrestorative sleep and fatigue are common symptoms of FM and OSA and may suggest related pathophysiology or co-morbidity that is yet to be diagnosed. This prospective randomized controlled clinical trial will enroll adult FM patients who screen positive for OSA by the STOP-Bang questionnaire. OSA will be confirmed by a laboratory polysomnography (PSG) study. After undergoing further baseline questionnaires and investigations, patients confirmed to have FM with moderate to severe OSA will be randomized to one of two different treatments: 1) Treatment for FM at the Chronic Pain Clinic together with Continuous Positive Airway Pressure (CPAP) devices for their OSA OR 2) Control group receiving treatment for FM at the Chronic Pain Clinic only.

DETAILED DESCRIPTION:
Sleep, pain and breathing have a complex multidimensional relationship. Pain disturbs sleep, poor sleep alters the perception of pain and sleep is a vulnerable state of breathing. The central system sensitization affecting the sensation of widespread pain in FM is due to a decrease in the neurophysiologic inhibition of perception of painful stimuli. This is caused by disturbed sleep. Rheumatic disease pathology can be understood in the light of the interference of cytokines and cellular immune functions with the sleeping/waking brain. Sleep disturbances such as unrefreshing sleep, difficulty falling asleep and frequent night awakenings have been reported by over 90% of FM patients. Sleep disturbances may be related to depression through pain and alteration of physical functioning. Depression and sleep disturbances have been proven to contribute to fatigue in FM patients. Although non-restorative sleep and fatigue are the most commonly reported symptoms by FM patients, the exact cause of these problems is not well understood. A study reported that 50% of the women with obstructive sleep apnea syndrome or upper airway resistance syndrome had chronic pain and more than 11 tender points. One case report has suggested OSA as a possible cause for FM. No studies have been conducted to demonstrate the effect of CPAP treatment on symptoms of FM syndrome in patients with OSA.

ELIGIBILITY:
Inclusion Criteria:

* Possesses cognitive and physical capability necessary to comprehend and complete the study questionnaires, as well as how to use CPAP machines.
* Be proficient in English, reading and comprehension at a Grade 6 level (patient or accompanying person).
* Be accessible for follow-up via interview appointments.
* Be able to provide informed consent.
* Has a Widespread Pain Index (WPI) score of ≥7 and Symptom Severity Score (SSS) of ≥5 OR a WPI 3-6 and SSS ≥9 according to 2010 American College of Rheumatology criteria for Fibromyalgia.
* Constant pain scores over the past 8 weeks.
* Newly diagnosed OSA patients with an AHI ≥15 OR AHI ≥5 on laboratory polysomnography with significant symptoms such as daytime sleepiness (Epworth Sleepiness Scale (ESS>10), or nocturnal symptoms (frequent nocturnal awakenings).

Exclusion Criteria:

* Conditions potentially interfering with comprehension and delivery of informed consent or unwillingness to provide consent.
* Psychiatric conditions interfering with necessary capability to comprehend and complete study questionnaires.
* Non-English speaking.
* Pregnant and lactating women.
* Uncorrectable coagulopathy interfering with phlebotomy.
* Contraindication to the application of a CPAP interface such as significant facial deformities, or skin lesions.
* History of drug or alcohol dependence or abuse within the last 3 months.
* History of primary pain disorders other than Fibromyalgia such as chronic pain disorder.
* History of primary sleep disorders associated with daytime sleepiness other than OSA, such as narcolepsy.
* Patients who do not meet the 2010 American College of Rheumatology Criteria for Fibromyalgia.
* Patients with previously diagnosed OSA who are already on CPAP before the initiation of the study.
* Patients receiving trigger point injections or intravenous lidocaine for pain treatment.
* Patients requiring an urgent sleep physician referral (within four weeks) due to serious medical conditions or safety critical-occupations according to the 2011 Canadian Thoracic Society (CTS) guidelines update e.g. unstable ischemic heart disease, recent cerebrovascular disease, congestive heart failure, refractory systemic hypertension, obstructive/restrictive lung disease, pulmonary hypertension, hypercapnic respiratory failure or pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Pain Score | 6 months
  Pain scores will measured on a Numerical Rating Scale (NRS) on the Brief Pain Inventory (BPI), reported at monthly intervals after allocation to a treatment group.

SECONDARY OUTCOMES:
Sleep quality | 6 months
  Sleep Quality will be measured via the Pittsburgh Sleep Quality Index (PSQI) and the Pain and Sleep Questionnaire (PSQ)
Sleepiness | 6 months
  Sleepiness will be measured via the Epworth Sleepiness Scale (ESS)
Quality of Life (QoL) | 6 months
  QoL will be measured via both the revised Fibromyalgia Impact Questionnaire (FIQR) and the Short Form 12 Health Survey (SF-12)
Inflammatory Marker | 6 months
  Measurement of serum levels of C-Reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Frances Chung, MBBS,FRCPC, Principal Investigator — University Health Network, Toronto Western Hospital and Women's College Hospital
Locations (2):
- Canada (2):
  - Women's College Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Yunus MB. Editorial review: an update on central sensitivity syndromes and the issues of nosology and psychobiology. Curr Rheumatol Rev. 2015;11(2):70-85. doi: 10.2174/157339711102150702112236. PMID 26138918
- [Background] Roizenblatt S, Neto NS, Tufik S. Sleep disorders and fibromyalgia. Curr Pain Headache Rep. 2011 Oct;15(5):347-57. doi: 10.1007/s11916-011-0213-3. PMID 21594765
- [Background] Fitzcharles MA, Ste-Marie PA, Goldenberg DL, Pereira JX, Abbey S, Choiniere M, Ko G, Moulin DE, Panopalis P, Proulx J, Shir Y; National Fibromyalgia Guideline Advisory Panel. 2012 Canadian Guidelines for the diagnosis and management of fibromyalgia syndrome: executive summary. Pain Res Manag. 2013 May-Jun;18(3):119-26. doi: 10.1155/2013/918216. PMID 23748251
- [Background] Peppard PE, Young T, Barnet JH, Palta M, Hagen EW, Hla KM. Increased prevalence of sleep-disordered breathing in adults. Am J Epidemiol. 2013 May 1;177(9):1006-14. doi: 10.1093/aje/kws342. Epub 2013 Apr 14. PMID 23589584
- [Background] Sepici V, Tosun A, Kokturk O. Obstructive sleep apnea syndrome as an uncommon cause of fibromyalgia: a case report. Rheumatol Int. 2007 Nov;28(1):69-71. doi: 10.1007/s00296-007-0375-9. Epub 2007 Jun 23. PMID 17589851
- [Background] Chung F, Subramanyam R, Liao P, Sasaki E, Shapiro C, Sun Y. High STOP-Bang score indicates a high probability of obstructive sleep apnoea. Br J Anaesth. 2012 May;108(5):768-75. doi: 10.1093/bja/aes022. Epub 2012 Mar 8. PMID 22401881
- [Result] Khalid I, Roehrs TA, Hudgel DW, Roth T. Continuous positive airway pressure in severe obstructive sleep apnea reduces pain sensitivity. Sleep. 2011 Dec 1;34(12):1687-91. doi: 10.5665/sleep.1436. PMID 22131606
- See also: The Official STOP-Bang Website — http://www.stopbang.ca